CLINICAL TRIAL: NCT04258267
Title: Which Factors Influence the Outcome After Anatomical and Reverse Shoulder Arthroplasty? A Prospective Longitudinal Study With Randomized Group Allocation, Towards Better Rehabilitation Strategies
Brief Title: Which Factors Influence the Outcome After Anatomical and Reverse Shoulder Arthroplasty?
Acronym: FINOSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Filip Struyf, Associate Professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19/48/559
Record Dates: First submitted 2020-01-16; First posted 2020-02-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Arthroplasty, Replacement, Shoulder
Keywords: "Influencing factors"; Rehabilitation; "Anatomical shoulder arthroplasty"; "Reverse shoulder arthroplasty"
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: Prospective longitudinal study with randomised group allocation, based on length of immobilization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The care provider and participant know the duration of the immobilization. The investigator and outcome assessor don't know the duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobilization (Experimental): Patients will be allowed to use their shoulder earlier. The immobilization period is shorter.
  Interventions: Procedure: Early mobilization
- Delayed mobilization (Experimental): The immobilization period is longer.
  Interventions: Procedure: Delayed mobilization

INTERVENTIONS:
Procedure: Early mobilization — Patients will wear an adduction sling to immobilize the shoulder during the first 4 weeks post-operative
  Arms: Early mobilization
Procedure: Delayed mobilization — Patients will wear an abduction sling to immobilize the shoulder during the first 4 weeks post-operative, followed by an adduction sling for 2 weeks.
  Arms: Delayed mobilization

SUMMARY:
The aim of this study is to investigate pre-, intra- and post-operative factors that influence post-operative outcome (shoulder pain, shoulder function and quality of life) after shoulder arthroplasty.

DETAILED DESCRIPTION:
The aim of this study is to investigate pre-, intra- and post-operative factors that influence post-operative outcome (shoulder pain, shoulder function and quality of life) after shoulder arthroplasty. Therefore, factors such as patient characteristics, indication for procedure, pre-operative shoulder pain, pre-operative shoulder function, patient expectations, psychosocial factors, lifestyle factors, length of immobilization and soft tissue integrity, are subject to study.

Secondary aims are to investigate:

1. the influences of early mobilization vs. delayed mobilization of the shoulder after shoulder arthroplasty on post-operative shoulder pain, shoulder function and quality of life.
2. the inter- and intrarater reliability of the test battery used in this project, in the shoulder arthroplasty population.
3. the inter- and intrarater reliability of the shoulder joint position sense (SJPS) test and the shoulder joint force sensation (SFS) test.
4. the routines of the orthopedic shoulder surgeons before, during and after performing a shoulder arthroplasty.
5. the routines of physiotherapists in the post-operative rehabilitation of patients with shoulder arthroplasty.
6. the associations between the Patient Reported Outcome Measures (PROMS) used in AZ Monica and the Constant Murley Score (CS), and the PROMS and the Visual Analogue Scale (VAS).

and to conduct a questionnaire - and assess its reliability - measuring the expectations of the shoulder arthroplasty patients.

In order to reach the aims of this project, a prospective longitudinal study with randomized group allocation will be carried out over 48 months with estimated starting point in January 2020 and finishing in January 2024.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women >= 18 years of age
* Scheduled for primary shoulder arthroplasty

Exclusion Criteria:

* Revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  There are 13 items, divided in two subscales: pain (5 items) and function (8 items). Each item is scored from 0 (no pain/no difficulty) to 10 (worst imaginable pain/so difficult it requires help) on a NPRS. The final score is a percentage derived from an average of the two subscales, where higher score means worse outcome.

SECONDARY OUTCOMES:
Shoulder pain | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  It is measured with the Visual Analogue Scale (VAS)
Shoulder function | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  It is measured with the Constant and Murley Score (CS)
Active ROM in shoulder abduction, anteflexion, internal rotation and external rotation | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  It is measured with a Gravity-V inclinometer. The unit of measures is degrees.
Shoulder muscle strength in anteflexion, internal rotation, external rotation and the lift-off movement | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  It is measured with a Handheld dynamometer. The unit of the measure is Newton.
Proprioception (joint position sense) | Measured pre-operatively, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  Inclinometer and laser pointer are used to measure joint position sense in degrees.
Proprioception (muscle force sensation) | Measured pre-operatively, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  A handheld dynamometer is used to measure muscle force sensation in Newton.
Patient related outcome measures (PROMS, EQ-D) | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  Questionnaire Lynxcare (Euro Quality of Life, 5 dimensions (EQ-5D)
Patient related outcome measures (PROMS, SST) | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  Questionnaire Lynxcare (Simple Shoulder Test (SST))
Patient related outcome measures (PROMS, NRS) | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  Questionnaire Lynxcare (Numeric Rating Scale (NRS))
Patient related outcome measures (PROMS, DASH) | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  Questionnaire Lynxcare (Disabilities of the Arm, Shoulder and Hand (DASH))
Quality of Life (SF-36) | Measured pre-operatively, 6 weeks post-operative, 12 weeks post-operative, 6 months postoperative, 12 months post-operative and 24 months post-operative
  It is a questionnaire to measure patient health, comprising mental health as well as physical health.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Monica, Deurne, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Claes A, De Mesel A, Struyf T, Verborgt O, Struyf F. Factors Influencing Outcome After Shoulder Arthroplasty (FINOSA Study): Protocol of a Prospective Longitudinal Study With Randomized Group Allocation. JMIR Res Protoc. 2024 Nov 18;13:e56522. doi: 10.2196/56522. PMID 39556824